CLINICAL TRIAL: NCT01575041
Title: Study on the Effects of Sodium and Potassium on Blood Pressure, Vascular Function and Renal Function in Untreated (pre)hypertensive Subjects
Brief Title: The Effects of Sodium and Potassium on Blood Pressure, Vascular Function and Renal Function
Acronym: KaNa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Principal Investigator, Marianne Geleijnse, Dr., Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: KaNa-trial
Record Dates: First submitted 2012-03-20; First posted 2012-04-10 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2012-08

CONDITIONS: Hypertension; Blood Pressure; Vascular Function; Renal Function
Keywords: sodium; salt; potassium; blood pressure; flow-mediated dilatation; endothelial function; renal function; controlled feeding study; dietary intervention
MeSH Terms: conditions — Hypertension | interventions — Sodium; Potassium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sodium (Active Comparator): For 4 weeks subjects will consume 3 grams of sodium by the intake of capsules on top of a low-sodium (2 grams of sodium), low-potassium (2 grams of potassium) diet
  Interventions: Dietary Supplement: Sodium
- Potassium (Active Comparator): For 4 weeks subjects will consume 3 grams of potassium by the intake of capsules on top of a low-sodium (2 grams of sodium), low-potassium (2 grams of potassium) diet.
  Interventions: Dietary Supplement: Sodium; Drug: Potassium
- Placebo (Placebo Comparator): For 4 weeks subjects will consume placebo capsules (content: cellulose) on top of a low-sodium low-potassium diet
  Interventions: Dietary Supplement: Sodium; Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Sodium — Sodium Chloride (provided by Microz, Geleen, Netherlands): 8 capsules per day which equals a sodium intake of 3 grams.
Drug: Potassium — Potassium Chloride (provided by Microz, Geleen, Netherlands): 8 capsules per day which equals a potassium intake of 3 grams.
  Arms: Potassium
Drug: Placebo — Placebo (cellulose, provided by Microz, Geleen, Netherlands): 8 capsules per day.
  Arms: Placebo

SUMMARY:
To determine the effect of (1) increased sodium intake and (2) increased potassium intake on blood pressure, vascular function and renal function in untreated (pre)hypertensive subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled cross-over feeding study.

ELIGIBILITY:
Inclusion Criteria:

* (Pre)hypertension, defined as office SBP: 130-159 mmHg;
* No use of antihypertensive, lipid-lowering, anticoagulant or other cardiovascular medication;
* Age at start of the ≥ 40 years;
* Apparently healthy:

  * No reported current or previous metabolic diseases
  * No history of cardiovascular diseases
  * No history of renal, liver or thyroid diseases
  * No history of gastrointestinal diseases
  * No diabetes mellitus
  * Fasting laboratory parameters within normal range: renal function (serum creatinine, ureum), liver function (ALAT, ASAT, ɣ-GT) and serum glucose.

Exclusion Criteria:

* Body mass index > 40 kg/m²;
* Smoking
* Secondary hypertension;
* Weight loss or weight gain of 5 kg or more during the last 2 months;
* Usage of non-steroidal anti-inflammatory drugs (aspirin, ibuprofen, naproxen) and not able or willing to stop taking them from at least 4 weeks prior to the study.
* Medical treatment that may affect blood pressure and not able (or willing) to stop taking them;
* Women taking oral contraceptives or estrogen replacement therapy
* Taking nutritional supplements and unwilling to discontinue;
* Women lactating, pregnant or intend to become pregnant during study;
* Reported dietary habits: medically prescribed diet, slimming diet;
* Reported alcohol consumption > 21 units/w (female subjects) or >28 units/w (male subjects);
* Unable or unwilling to consume one meal every workday at the university, or to consume the prescribed study diet for 13 weeks;
* Problems with consuming the supplements or following the study guidelines;
* Unwilling to undergo home or office blood pressure measurements;
* Recent blood donation i.e. 1 month (male subjects) or 2 months (female subjects) prior to the study and planned donation during the study period;
* Reported intense sporting activities > 10 h/w;
* Not agreeing to be informed about unexpected and medically relevant personal test-results
* Participation in another biomedical trial less than 2 months before the start of the study or at the same time;
* No informed consent signed.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in Endothelium-dependent flow-mediated dilation comparing (1) high sodium, low potassium intake and (2) low sodium, high potassium intake with low sodium, low potassium intake. | Baseline at week 1 (t=0). After intervention period 1 at week 5 (t=1). After intervention period 2 at week 9 (t=2). After intervention period 3 at week 13 (t=3)
  Ultra-sonography (brachial artery) + Picus system

SECONDARY OUTCOMES:
Change in blood pressure comparing (1) high sodium, low potassium intake and (2) low sodium, high potassium intake with low sodium, low potassium intake. | Screening. Baseline at week 1 (t=0). After intervention period 1 at week 5 (t=1). After intervention period 2 at week 9 (t=2). After intervention period 3 at week 13 (t=3)
  Includes:
  Office BP (Dinamap, 4 consecutive measurements with 2-min intervals) ABPM (Spacelab; 1x24h, at baseline, week 5, week 9, week 13)
Change in Pulse Wave Velocity comparing (1) high sodium, low potassium intake and (2) low sodium, high potassium intake with low sodium, low potassium intake. | Baseline at week 1 (t=0). After intervention period 1 at week 5 (t=1). After intervention period 2 at week 9 (t=2). After intervention period 3 at week 13 (t=3)
  Device: SphygmoCor (tonometry)
  Parameters: Pulse Wave Velocity and at baseline, week 5, week 9 and week 13
Change in vasomotion comparing (1) high sodium, low potassium intake and (2) low sodium, high potassium intake with low sodium, low potassium intake. | Baseline at week 1 (t=0). After intervention period 1 at week 5 (t=1). After intervention period 2 at week 9 (t=2). After intervention period 3 at week 13 (t=3)
  Device: PeriFlux 5000 (Perimed, Sweden0
Change in Biomarkers of endothelial function comparing (1) high sodium, low potassium intake and (2) low sodium, high potassium intake with low sodium, low potassium intake. | Baseline at week 1 (t=0). After intervention period 1 at week 5 (t=1). After intervention period 2 at week 9 (t=2). After intervention period 3 at week 13 (t=3)
  Plasma analysis of endothelin-1, ADMA, MCP-1, sVCAM-1, sICAM-1, sE-selectin, sTM, CRP, SAA, IL-6, IL-8, TNF-α, vWF, nitric oxide
Change in renal function comparing (1) high sodium, low potassium intake and (2) low sodium, high potassium intake with low sodium, low potassium intake. | Screening. Baseline at week 1 (t=0). After intervention period 1 at week 5 (t=1). After intervention period 2 at week 9 (t=2). After intervention period 3 at week 13 (t=3)
  eGFR, serum creatinine (at screening also used as safety parameter)
Change in cardiovascular parameters in plasma comparing (1) high sodium, low potassium intake and (2) low sodium, high potassium intake with low sodium, low potassium intake. | Screening. Baseline at week 1 (t=0). After intervention period 1 at week 5 (t=1). After intervention period 2 at week 9 (t=2). After intervention period 3 at week 13 (t=3)
  Total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides, insulin and glucose (at screening also used as safety parameter)
Liver function parameters | Screening. Baseline at week 1 (t=0). After intervention period 1 at week 5 (t=1). After intervention period 2 at week 9 (t=2). After intervention period 3 at week 13 (t=3)
  Montoring liver function parameters for safety: includes ALAT, ASAT and ɣ-GT
24-hour urinary mineral excretions | Screening. Baseline at week 1 (t=0). After intervention period 1 at week 5 (t=1). After intervention period 2 at week 9 (t=2). After intervention period 3 at week 13 (t=3)
  Sodium and potassium (as compliance markers)
24-hour excretion of protein, albumin and creatinine | Screening. Baseline at week 1 (t=0). After intervention period 1 at week 5 (t=1). After intervention period 2 at week 9 (t=2). After intervention period 3 at week 13 (t=3)
  In addition, protein is assessed in spot urine during screening using a dipstick test
Adverse events | Every day
  Patient diary for occasions of illness, hospitalizations, medication use and other information on potential side effects
Anthropometric measurements | Screening. Baseline at week 1 (t=0). After intervention period 1 at week 5 (t=1). After intervention period 2 at week 9 (t=2). After intervention period 3 at week 13 (t=3)
  Body weight (weekly), height (only at baseline), waist circumference (baseline and every 4 weeks)
Heart rate | Screening. Baseline at week 1 (t=0). After intervention period 1 at week 5 (t=1). After intervention period 2 at week 9 (t=2). After intervention period 3 at week 13 (t=3)
  Dinamap, 4 consecutive measurements with 2-min intervals
Food frequency questionnaire | Screening
Change in Pulse Wave Analysis comparing (1) high sodium, low potassium intake and (2) low sodium, high potassium intake with low sodium, low potassium intake. | Baseline at week 1 (t=0). After intervention period 1 at week 5 (t=1). After intervention period 2 at week 9 (t=2). After intervention period 3 at week 13 (t=3)
  Device: SphygmoCor (tonometry)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna M Geleijnse, PhD, Principal Investigator — Wageningen University, Division of Human Nutrition
Locations (1):
- Wageningen University, Wageningen, Netherlands

REFERENCES:
- [Derived] Humalda JK, Yeung SMH, Geleijnse JM, Gijsbers L, Riphagen IJ, Hoorn EJ, Rotmans JI, Vogt L, Navis G, Bakker SJL, de Borst MH. Effects of Potassium or Sodium Supplementation on Mineral Homeostasis: A Controlled Dietary Intervention Study. J Clin Endocrinol Metab. 2020 Sep 1;105(9):e3246-56. doi: 10.1210/clinem/dgaa359. PMID 32506135
- See also: Website of the Top Institute Food and Nutrition, Wageningen, The Netherlands — http://www.tifn.nl